CLINICAL TRIAL: NCT04182750
Title: Promoting Safe Medication Use in Pregnancy in the Era of Real-World Data - The SafeStart Study
Acronym: SafeStart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hedvig Marie Egeland Nordeng (Other)
Responsible Party: Sponsor-Investigator, Hedvig Marie Egeland Nordeng, Professor, University of Oslo
Organization: University of Oslo (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SafeStart
Record Dates: First submitted 2019-11-22; First posted 2019-12-02 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Pregnancy Early; Emesis; Medication Adherence
MeSH Terms: conditions — Vomiting; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Pharmacist consultation in early pregnancy (gestation week <12)
  Interventions: Other: Pharmacist consultation
- Control group (No Intervention): Standard care.

INTERVENTIONS:
Other: Pharmacist consultation — The intervention is a patient-centered consultation that will last about 15 minutes. The intervention is defined as "A planned, individualized, and structured conversation with the purpose to relieve pregnant women for any concern and answer questions she may have regarding self-care ailments and medication use in pregnancy". Specifically, the consultation will:
  * Answer any questions the participants may have within pharmaceutical care.
  * Improve pregnant women's understanding of common pregnancy-related ailments and hence contribute to better management of the ailments.
  * Raise awareness, provide confidence, and give information about safe medications options in pregnancy
  * Focus on preventative measures for NVP.
  * Contribute to better adherence for needed/chronic medication throughout the pregnancy.
  The pharmacists will beforehand have access to the women´s answers from the baseline questionnaire Q1, including information about her medical conditions and medication use.
  Arms: Intervention group

SUMMARY:
The background for this project is the growing concern about women's use of medications during pregnancy. Several studies have shown that up to 80% of all pregnant women use at least one medication during pregnancy, most commonly prescription-free medications for pregnancy-related ailments. Despite the frequent use of medications during pregnancy pregnant women tend to overestimate the teratogenic risk of medications - often resulting in unfound anxiety, non-adherence to needed medication, use of herbal "natural" medications, and in the worst case, termination of otherwise wanted pregnancies. Specifically, the investigators have found that ailments such as nausea and vomiting in pregnancy (NVP), often are mismanaged, resulting in profound impacts on the women´s quality of life, but are often being neglected by healthcare personnel.

The objective of this project is to investigate whether a pharmacist consultation provided in early pregnancy can result in optimized management of pregnancy-related ailment, a higher quality of life and reduce sick leave among pregnant women. The investigators will capitalize on the existence of a unique personal identification number allocated to every citizen in Norway and link the self-reported data generated in the intervention study to five national health registries. As even mild NVP has been shown to have a huge impact on pregnant women's quality of life, the investigators will specifically focus on preventative measures for NVP.

The investigators main hypothesis is:

"A pharmacist intervention focusing on safe medication use and in early pregnancy can reduce sick leave days and rates, enhance adherence, promote better management of common pregnancy-related ailments (especially NVP), and improve pregnant women's quality of life"

The investigators will include all pregnant women in pregnancy weeks <12. Pregnant women under the age of 18, women who do not understand Norwegian and women for some other reason are unable to sign the consent form will be excluded. Women eligible for inclusion will be allocated to either the intervention group or the control group. Participants in the intervention group will be directed to the nearest study pharmacy for the intervention. The proposed study intervention is to be applied and carried out in the community pharmacy. Approximately 10-15 community pharmacists across the country will be involved. If the distance to a study pharmacy is too far for a physical meeting, the intervention will be performed over the telephone; otherwise, the private information room in the pharmacies will be utilized.

All pharmacists involved in the study will be specifically trained to perform the consultation. They will complete several e-learning modules on pharmacotherapy in pregnancy and attend a full-day training work-shop focusing on communication skills led by experienced clinical pharmacists.

Data will be collected by four online questionnaires, one at baseline in the first trimester, one during the second trimester, one during the third trimester, and the last one in the post-partum period. Participants in the intervention group will, in addition, complete a satisfaction questionnaire right after the completion of the consultation. All questionnaires will be distributed to the participants by email. Data about the participants will, in addition, be collected from five national registries; National Sick Leave Database (Forløpsdatabasen Trygd), The Norwegian Patient Registry, The Norwegian Prescription Database, The Medical Birth Registry of Norway, and the Municipality Patient and User Registry (Kommunalt Bruker- og Pasientregister). These data will be linked to the self-reported data (by the unique identification number of every citizen in Norway) collected during the intervention study.

An economic evaluation will be done to assess the cost-effectiveness of the intervention.

All study pharmacists involved in the study will be invited to participate in a qualitative interview to share their experience and opinions regarding the pharmacist intervention.

Participants enrolled in the intervention study will be invited to a qualitative interview to share their inputs and opinions on what a mobile application for self-management and an online patient-centered decision support tool for NVP should include.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant in the first trimester (< gestational week 12)
* Speaks/understand Norwegian

Exclusion Criteria:

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 369 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Change in quality of life between the first and second trimester | Change in quality of life between the first (gestation week < 12) and second trimester (between gestation week 17 and 25)
  Quality of life measured by the Quality of Life Scale (QOLS) which ranges from 16 to 112, where higher score indicates better quality of life
Sick leave during the first trimester | Up to weeks 12
  Self-reported sick leave rate and days and as recorded in the national registry (Forløpsdatabasen Trygd) during the first trimester (up to weeks 12)
Sick leave during the second trimester | Between weeks 13 and 28
  Self-reported sick leave rate and days and as recorded in the national registry (Forløpsdatabasen Trygd) during the second trimester (between weeks 13 and 28)
Sick leave during the third trimester | Between weeks 29 and delivery
  Self-reported sick leave rate and days and as recorded in the national registry (Forløpsdatabasen Trygd) during the third trimester (between weeks 19 and delivery)
Sick leave in the post-partum period | From delivery and up to three months post-partum
  Self-reported sick leave rate and days and as recorded in the national registry (Forløpsdatabasen Trygd) from delivery and up to three months post-partum
Utilization of health care services during the first trimester | Up to weeks 12
  Self-reported number of visits and as recorded in the Norwegian Patient Registry during the first trimester (up to weeks 12)
Utilization of health care services during the second trimester | Between weeks 13 and 28
  Self-reported number of visits and as recorded in the Norwegian Patient Registry during the second trimester (between weeks 13 and 28)
Utilization of health care services during the third trimester | Between weeks 29 and delivery
  Self-reported number of visits and as recorded in the Norwegian Patient Registry during the third trimester (between weeks 29 and delivery)
Utilization of health care services in the post-partum period | From delivery and up to three months post-partum.
  Self-reported number of visits and as recorded in the Norwegian Patient Registry from delivery and up to three months post-partum
Use of medications during the first trimester | Up to weeks 12
  Self-reported medication use and as recorded in the Norwegian Prescription Database during the first trimester (up to weeks 12)
Use of medications during the second trimester | Between weeks 13 and 28
  Self-reported medication use and as recorded in the Norwegian Prescription Database during the second trimester (between weeks 13 and 28)
Use of medications during the third trimester | Between weeks 29 and delivery
  Self-reported medication use and as recorded in the Norwegian Prescription Database during the third trimester (between weeks 29 and delivery)
Use of medications in the post-partum period | From delivery and and up to three months post-partum.
  Self-reported medication use and as recorded in the Norwegian Prescription Database from delivery and up to three months post-partum
Quality-Adjusted-Life-Years (QALY) during the first trimester | Up to weeks 12
  Participants' Quality-Adjusted-Life-Years (QALYs) measured by the EuroQoL health-related quality of life instrument (EQ-5D-5L) during the first trimester. The EQ-5D-5L state will be converted to an index value (based on the most appropriate weights available for the Norwegian population) and further to QALYs. QALYs ranges from 0 (death) to 1 (full or optimal health).
Quality-Adjusted-Life-Years (QALY) during the second trimester | Between weeks 13 and 28
  Participants' Quality-Adjusted-Life-Years (QALY) measured by the EuroQoL health-related quality of life instrument (EQ-5D-5L) during the second trimester. The EQ-5D-5L state will be converted to an index value (based on the most appropriate weights available for the Norwegian population) and further to QALYs. QALYs ranges from 0 (death) to 1 (full or optimal health).
Quality-Adjusted-Life-Years (QALY) during the third trimester | Between weeks 29 and delivery
  Participants' Quality-Adjusted-Life-Years (QALY) measured by the EuroQoL health-related quality of life instrument (EQ-5D-5L) during the third trimester. The EQ-5D-5L state will be converted to an index value (based on the most appropriate weights available for the Norwegian population) and further to QALYs. QALYs ranges from 0 (death) to 1 (full or optimal health).
Quality-Adjusted-Life-Years (QALY) in the post-partum period | Between delivery and up to three months post-partum
  Participants' Quality-Adjusted-Life-Years (QALY) measured by the EuroQoL health-related quality of life instrument (EQ-5D-5L) from delivery and up to three months post-partum. The EQ-5D-5L state will be converted to an index value (based on the most appropriate weights available for the Norwegian population) and further to QALYs. QALYs ranges from 0 (death) to 1 (full or optimal health).
Economic evaluation of the intervention | After intervention completion (up to weeks 12)
  All costs related to performing the intervention, reported by the study pharmacists
Economic evaluation of the intervention | 1 year
  Cost related to sick leave as recorded in the national registry Forløpsdatabasen Trygd during pregnancy and up to three months post-partum

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Schultz, Study Director — Department of Pharmacy, University of Oslo
Locations (1):
- Department of Pharmacy, University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available because of data protection regulation.

REFERENCES:
- [Derived] Ngo E, Truong MB, Nordeng H. Impact of a primary care pharmacist consultations on pregnant women's medication use: the SafeStart intervention study linked to a national prescription database. Int J Clin Pharm. 2023 Aug;45(4):893-902. doi: 10.1007/s11096-023-01577-x. Epub 2023 May 8. PMID 37156960
- [Derived] Truong MB, Ngo E, Ariansen H, Tsuyuki RT, Nordeng H. The effect of a pharmacist consultation on pregnant women's quality of life with a special focus on nausea and vomiting: an intervention study. BMC Pregnancy Childbirth. 2020 Dec 9;20(1):766. doi: 10.1186/s12884-020-03472-z. PMID 33298010